CLINICAL TRIAL: NCT01471418
Title: Investigation of the Use of Positron Emission Tomography With 18F-FDG PET/CT for the Diagnosis of Synovitis in the Temporomandibular Joint
Brief Title: The Use of PET/CT to Evaluate Synovitis in the Temporomandibular Joint (TMJ)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 29-Apr-14 UPENN IRB granted approval to close study due to lack of funding
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 813671
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Temporomandibular Joint; Conservative Treatment Therapy
Keywords: TMJ; orofacial pain; synovitis; arthroscopy
MeSH Terms: conditions — Facial Pain; Synovitis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Disease population (Experimental)
  Interventions: Drug: PET/CT with 18-FDG

INTERVENTIONS:
Drug: PET/CT with 18-FDG — FDG uptake

SUMMARY:
Temporomandibular joint disorders (TMD) are a common musculoskeletal problem with an estimated 40-75 percent of the population reporting at least one sign. Up to fifteen percent of the patients who seek care for one of these conditions, will go on to develop chronic pain. The two most common TMD conditions include myofascial pain disorder and internal derangement of the Temporomandibular Joint (TMJ). These two conditions have similar clinical presentations, making an accurate diagnosis difficult. Currently, there is no accurate exam or test to differentiate between these two conditions.

Internal derangement of the TMJ is a condition with disk displacement, pain, and dysfunction, which may progress to localized osteoarthritis. Fortunately, this condition is self-limiting for the majority of the patients afflicted, with a small minority progressing to advanced joint destruction, disability and chronic pain.18 Currently there are no prognostic indicators to identify these individuals. There are three hypothesis of degenerative TMJ disease, they include: direct mechanical trauma, hypoxia reperfusion injuries, and neurogenic inflammation. All involve parafunctional habits such as clenching or grinding by the patient and a low-grade inflammatory response/synovitis. 18-fluorodeoxyglucose (18-FDG), a radioisotope used with positron emission tomography (PET) and paired with a CT scan (PET/CT), may have a role in imaging inflammation in arthritis as recently demonstrated in several pilot studies involving osteoarthritis of the knee and shoulder. 18-FDG accumulates in areas of increased metabolism, particularly activated leukocytes, as measured by increased standardized uptake value.2 PET/CT offers the unique advantage of showing active disease before anatomic damage is evident. Our hypothesis is that there is an increased uptake of 18-FDG on PET/CT in synovitis of the TMJ.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, pilot study to evaluate the ability of PET/CT with FDG to detect synovitis of the temporomandibular joint. Patients presenting to the Department of Oral and Maxillofacial Surgery at the Hospital of the University of Pennsylvania with symptomatic internal derangement of the temporomandibular joint requiring arthroscopy will be compared to control subjects. Key inclusion criteria include any individual found to have a primary diagnosis of internal derangement of the temporomandibular joint requiring arthroscopy as determined by the treating physician. All patients will have failed a trial period of "conservative treatment therapy" including occlusal splint therapy, NSAIDs, or muscle relaxants for a period no less than eight weeks. Exclusion criteria will include patients not medically stable to undergo arthroscopy under general anesthesia, patients with overlying infection of the skin, patients with conditions other than internal derangement causing temporomandibular pain or dysfunction.

Once a patient has been identified as eligible for the study, the treating physician will contact a member of the study team. Each participating patient will undergo a standardized exam, the research diagnostic criteria for TMD (RDC/TMD). A member of the research team, from the department of oral medicine, will administer this exam. This standardized exam has been previously validated in the literature, and each member of the research team will undergo training and calibration prior to administering the RDC/TMD. This exam will be performed on the day of the arthroscopy. In addition, each patient will be given a Wilkes score, based on the Wilkes classification of internal derangement.36 The patient will then undergo arthroscopy of the temporomandibular joint as per the treating physician. TMJ arthroscopy includes: a small incision in front of the ear, introduction of an arthroscope and irrigation needle into the joint space, irrigation of fluid, and at the discretion of the treating physician may include the lysis of adhesion and the introduction of medication into the joint. At the time of the procedure, the synovitis score will be determined based on an eleven point synovitis scale as described by Murakami, with zero being absence of synovial inflammation. This scoring is bone by observation, and is typically include in the arthroscopy procedure for diagnosis. The patient will also be given a binomial score of presence or absence of synovitis. A representative photograph will be obtained of the patient's joint during arthroscopy, as is routinely done during this procedures.

Prior to the procedure, the patients will have undergone a PET/CT scan to evaluate the TMJ. This radiographic exam will be limited to the head and neck region in order to minimize radiation exposure. The radiologists reading the study will be blinded to the results of the clinical exam and condition. The results of the PET/CT study will be given as a binomial score of positive or negative and given a continuous score based on uptake relative to the unaffected joint.

Control subjects will undergo the RDC/TMD standardized exam prior to the radiographic study, and only have the PET/CT performed, with no subsequent intervention. These patients will be aged matched to the treatment subjects. This information will then be utilized to determine the utility of PET/CT in the detection of synovitis of the temporomandibular joint.

ELIGIBILITY:
Inclusion Criteria:

* Key inclusion criteria include any individual found to have a primary diagnosis of internal derangement of the temporomandibular joint requiring arthroscopy as determined by the treating physician.
* All patients will have failed a trial period of "conservative treatment therapy" including occlusal splint therapy, NSAIDs, or muscle relaxants for a period no less than eight weeks, as per standard of care.
* All patients will be between the ages of 18 and 70.

Exclusion Criteria:

* Exclusion criteria will include patients not medically stable to undergo arthroscopy under general anesthesia, patients with overlying infection of the skin, uncontrolled diabetes, patients with bilateral TMJ internal derangement, pregnancy, and patients with conditions other than internal derangement causing temporomandibular pain or dysfunction.
* Patients less than 18 or greater than 70 years of age will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable will be the presence or absence of 18F-FDG uptake on positron emission tomography combined with computed tomography (CT) of the temporomandibular joint. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States